CLINICAL TRIAL: NCT04879199
Title: Stop Tip-toeing Around Toe-walking: Towards a Better Understanding and More Effective Treatment of Toe-walkers With Cerebral Palsy
Brief Title: Stop Tip-toeing Around Toe-walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-00435; ks21Viehweger
Record Dates: First submitted 2021-05-03; First posted 2021-05-10 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Spastic Cerebral Palsy (sCP)
Keywords: tip-toeing; toe-walking; gait cycle; heel-strike; Static stability; Dynamic stability; Virtual Reality; Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Cross sectional, age-matched-controlled and monocentric study with an exploratory approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Typically Developing (TD) children (Experimental): Static stability and Dynamic stability measurement in children with: 1) between the age of 7 and 18 years, 2) who are typically developing, 3) able to stand and walk alone without using assistance or assistive devices, 4) able to place their feet flat on the force platforms, and 5) with enough German language skills to follow the instructions.
  Interventions: Diagnostic Test: Static stability measurement; Diagnostic Test: Dynamic stability measurement
- Spastic Cerebral Palsy (sCP) children (Experimental): Static stability and Dynamic stability measurement in children with: 1) between the age of 7 and 18 years, 2) with the diagnosis of spastic CP or CP similar (both unilateral and bilateral), functionally classified level I or II according to the Gross Motor Function Classification System (GMFCS) [98], 3) being able to stand and walk alone without assistance or assistive devices, 4) able to place their feet flat on the force platforms, and 5) with enough German language skills to follow the instructions.
  Interventions: Diagnostic Test: Static stability measurement; Diagnostic Test: Dynamic stability measurement

INTERVENTIONS:
Diagnostic Test: Static stability measurement — The child stands barefoot on dual force platforms in two (CP: three) different conditions: barefoot and with shoes (CP: and with orthosis). Each condition is recorded three times each lasting for 30s, and 30s rest between them. Both conditions are recorded with and without wearing a headset. The order of conditions (within each Virtual Reality ("VR)-condition") is randomized. For each condition, the child rests in a comfortable position for 20s with the heels on the same level and arms hanging at their sides. Between both "VR-conditions", the child rests for 120 s.
Diagnostic Test: Dynamic stability measurement — The child walks at their normal walking speed on a 10-m walkway in two (CP: three) different conditions: barefoot and with shoes (CP: and with orthosis). For each condition, at least six error-free trials are recorded. Errors in data may occur due to hidden or lost markers during walking or software interruptions. Both conditions are recorded with and without wearing a headset. The order of conditions (within each "VR-condition") is randomized.

SUMMARY:
The purpose of this study is to explore the interplay among nervous-, musculoskeletal-, and psychological systems and how they impact toe-walking behavior, and vice versa.

Sub-Project 1 is to analyze the feasibility of the developed virtual reality (VR) environment, in 10 TD and sCP children respectively. It is assess the effects of VR immersion on predefined static and dynamic stability parameters.

Sub-Project 2: After adjustments have been made following Sub-Project 1 regarding the study procedure, technical factors or the parameters of interest etc., the optimized study procedure is implemented in Sub-Project 2 (20 to 25 TD will be included).

Sub-Project 3: After adjustments have been made following Sub-Project 1 regarding the study procedure, technical factors or the parameters of interest etc., the optimized study procedure is implemented in Sub-Project3 (20 to 25 sCP will be included)

DETAILED DESCRIPTION:
The interplay between the nervous-, musculoskeletal-, and psychological systems and their impact on resulting walking patterns are poorly understood. Children that toe-walk often show poorer levels of static and dynamic stability, leading to a lower quality of life compared to typically develop-ing children (TD). Current research suggests multifactorial adaptations in central and/or peripheral nervous as well as the musculoskeletal system contribute to and result from toe-walk-ing. The purpose of this study is to explore the interplay among nervous-, musculoskeletal-, and psychological systems and how they impact toe-walking behavior, and vice versa. The effect of psychological factors (via the use of a custom-designed virtual reality environment) on static vs. dynamic stability, motor control, coordination (indirect assessment of central nervous system function) as well as reflex control (Hoffmann-reflex, H-reflex, performance of peripheral nervous system) is investigated.

ELIGIBILITY:
Inclusion Criteria for TD children:

* between the age of 7 and 18 years
* who are typically developing
* able to stand and walk alone without using assistance or assistive devices
* able to place their feet flat on the force platforms
* with enough German language skills to follow the instructions

Inclusion Criteria for sCP children:

* between the age of 7 and 18 years
* with the diagnosis of spastic CP or CP similar (both unilateral and bilateral), functionally classified level I or II according to the Gross Motor Function Classification System (GMFCS)
* being able to stand and walk alone without assistance or assistive devices
* able to place their feet flat on the force platforms
* with enough German language skills to follow the instructions

Exclusion Criteria for TD children:

* severe visual, cognitive, or auditory impairments that would interfere with the study instructions and the VR immersion
* any vestibular problems (e.g. severe motion sickness)
* history of epilepsy, pace-marker or/and electrical pumps (due to possible interference with electrical stimulation)
* prior experience of VR to ensure a comparable baseline between subjects

Exclusion Criteria for sCP children:

* severe visual, cognitive, or auditory impairments that would interfere with the study instructions and the VR immersion
* severe knee flexion gait (>45°)
* walking capacity <50m
* botulinum toxin type A treatment (past 6 months)
* orthopedic surgery of upper or lower extremities (past 12 months)
* any vestibular problems (e.g. severe motion sickness or dizziness)
* history of epilepsy, pace-marker or/and electrical pumps (due to possible interference with electrical stimulation)
* prior experience of VR as they may already be adapted to VR.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Static stability assessed by Center of Pressure (COP) shifts in anterior-posterior and mediolateral directions under each limb | one time assessment at baseline (complete baseline assessments up to 3 hours)
  COP shifts in anterior-posterior and mediolateral directions under each limb are assessed via the use of two force plates embedded in the floor (Kistler Instrumente AG, Winterthur, Switzerland, sample rate 1500 Hz) (mean value of three repetitions)
Static stability assessed by Visual Analogue Scale (VAS) | one time assessment at baseline (complete baseline assessments up to 3 hours)
  Self-perceived degree of safety during walking in the VR environment will be assessed using a Visual Analogue Scale (VAS) ranging from 0 ("feeling completely safe") to 10 ("feeling completely unsafe")
Static stability assessed by Ratio between H-reflex and M-wave amplitude | one time assessment at baseline (complete baseline assessments up to 3 hours)
  Ratio between H-reflex and M-wave amplitude, measured through soleus muscle in affected side of hemiplegic sCP and in none-dominant side for diplegic CP and TD (recruitment curve of the H-reflex and the M-wave of the Soleus elicited by stimulating the tibial nerve while standing)
Dynamic stability assessed by COP shifts in combination with base of support trajectory | one time assessment at baseline (complete baseline assessments up to 3 hours)
  COP shifts in combination with base of support trajectory assessed via the use of four force plates embedded in the floor (mean value of three repetitions)
Dynamic stability assessed by number of muscle synergies | one time assessment at baseline (complete baseline assessments up to 3 hours)
  Number of muscle synergies assessed via the use of a sixteen-channel surface electromyography system
Dynamic stability assessed by interlimb coordination | one time assessment at baseline (complete baseline assessments up to 3 hours)
  Interlimb coordination will be calculated by using kinematic data from lower and upper extremities
Dynamic stability assessed by Self-perceived degree of safety during walking in the VR environment using a Visual Analogue Scale (VAS) | one time assessment at baseline (complete baseline assessments up to 3 hours)
  Dynamic stability assessed by Self-perceived degree of safety during walking in the VR environment using a Visual Analogue Scale (VAS) ranging from 0 ("feeling completely safe") to 10 ("feeling completely unsafe")

SECONDARY OUTCOMES:
Dynamic stability measurement assessed by kinematic data of upper & lower extremities (joint angles in degree) | one time assessment at baseline (complete baseline assessments up to 3 hours)
  Dynamic stability measurement assessed by kinematic data of upper & lower extremities (joint angles in degree)
Dynamic stability measurement assessed by spatiotemporal parameters: walking speed (normalized to leg length) [m/(s*mm)] | one time assessment at baseline (complete baseline assessments up to 3 hours)
  Dynamic stability measurement assessed by spatiotemporal parameters: walking speed (normalized to leg length) [m/(s*mm)]
Dynamic stability measurement assessed by spatiotemporal parameters: stride width [s] | one time assessment at baseline (complete baseline assessments up to 3 hours)
  Dynamic stability measurement assessed by spatiotemporal parameters: stride width [s]
Dynamic stability measurement assessed by spatiotemporal parameters: double support time [s] | one time assessment at baseline (complete baseline assessments up to 3 hours)
  Dynamic stability measurement assessed by spatiotemporal parameters: double support time [s]
Dynamic stability measurement assessed by spatiotemporal parameters: cadence [steps/min] | one time assessment at baseline (complete baseline assessments up to 3 hours)
  Dynamic stability measurement assessed by spatiotemporal parameters: cadence [steps/min]
Dynamic stability measurement assessed by spatiotemporal parameters: step length [m] | one time assessment at baseline (complete baseline assessments up to 3 hours)
  Dynamic stability measurement assessed by spatiotemporal parameters: step length [m]

CONTACTS AND LOCATIONS:
Overall Officials: Heide Elke Viehweger, Prof. Dr. med., Principal Investigator — University Children's Hospital Basel, Neuroorthopedics I Human Locomotion Research
Locations (1):
- University Children's Hospital Basel, Neuroorthopedics I Human Locomotion Research, Basel, Switzerland